CLINICAL TRIAL: NCT01605630
Title: Family Cancer Literacy to Promote Mammography Screening Among Navajo Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Christi Patten, Professor of Psychology, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-004328; R21CA152433 (NIH)
Record Dates: First submitted 2012-05-07; First posted 2012-05-25 (Estimated); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Family-based cancer literacy intervention (Experimental)
  Interventions: Behavioral: Family-based family cancer literacy intervention
- Control (Active Comparator): Standard of care
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Family-based family cancer literacy intervention — family based counseling and materials provided in navajo/english including digital stories
  Arms: Family-based cancer literacy intervention
Behavioral: Control — standard of care
  Arms: Control

SUMMARY:
The no show rate for mammography screening is high among Navajo women. One barrier to preventive screening is a lack of cancer literacy including low knowledge and cultural attitudes (e.g., fatalism) about screening. The investigators will examine the potential feasibility and acceptability of a cancer literacy intervention for families of Navajo women who have no showed for three consecutive times to mammography screening who have never or rarely been screened in the past.

DETAILED DESCRIPTION:
This proposal describes a community-based participatory research study to develop and pilot test a new behavioral intervention to promote mammography screening among Navajo women. From a public health perspective, the intervention has the potential to reach many Navajo women, as 80% of women scheduled for mammography appointments do not follow through. These women (over 1,500 each year) are referred to the Nation Breast and Cervical Cancer Prevention Program (NNBCCPP). A key barrier toward implementing cancer prevention and control efforts in the Navajo community is a lack of cancer literacy or cultural and conceptual knowledge regarding cancer. Other barriers to screening are fear of cancer, stigma of cancer (even talking about cancer) often experienced by the patient, family and community, and lack of knowledge about the etiology of cancer and importance of early detection. Therefore, communication about cancer is impeded within Navajo families and the community.

This proposal builds on our successful partnership and collaboration with Diné College (the Navajo tribal college). The proposed study is designed to assess the feasibility and potential efficacy of a cancer-literacy focused, family-based intervention on completion of mammography screening for Navajo women. The intervention will include culturally and linguistically appropriate educational materials about cancer (e.g., the Navajo Cancer Glossary). The project will be implemented in two phases. During Phase 1, the investigators will develop the family cancer literacy intervention with feedback from our community advisory committee. In addition, the Cancer Literacy Measure will be adapted for Navajo women through focus groups and individual interviews. Phase 2 will consist of a formative evaluation of the intervention. The NNBCCPP patient and a female family member will be randomly assigned in pairs to the control condition (existing NNBCCPP health education services, N=40 pairs) or to receive these health education services plus the family cancer literacy intervention (N=40 pairs). The investigators will assess the intervention's feasibility and acceptability as indicated by the recruitment and retention rates and qualitative ratings of treatment acceptability. In addition, the investigators will examine the effect of the intervention compared with the control group on the proportion of women who complete mammography screening at 3-month follow-up documented by NNBCCPP records. The investigators will also examine changes in Cancer Literacy Measure scores from baseline to 3-month follow-up among both patients and family members. The investigators expect that as a result of this project, the investigators will have developed a replicable, feasible, and acceptable intervention, the efficacy of which can be tested in future large-scale randomized clinical trials. In addition, the adapted Cancer Literacy Measure could be used in future cancer prevention and control projects within the Navajo Nation. The overall objective is to reduce breast cancer morbidity and mortality among Navajo women.

ELIGIBILITY:
Inclusion Criteria:

In Phase 1, we will recruit 17 Navajo women for individual interviews (n=5) and focus groups (n=12) to adapt our measures. Eligibility criteria are:

1. aged 40 years or older and
2. provides written informed consent. We chose to develop our measures based on feedback from the general community of women who are screening eligible instead of matching the inclusion/exclusion criteria to that used in the formative evaluation of the intervention (Phase 2). This will enhance our ability to use the Cancer Literacy Measure and other assessments in subsequent breast cancer prevention and control studies.

In Phase 2, we will recruit a total of 40 patient-family member pairs. To be eligible for the study, the NNBCCPP patient must:

1. be aged 40 years or older,
2. provide written informed consent,
3. be referred to the NNBCCPP as a "no-show" for mammography screening after three scheduling attempts,
4. have no prior history of mammography screening,
5. have no prior history of breast cancer, and
6. can identify a female family member or other individual who resides in or near the home who could participate in the project.

In addition, the family member must:

1. be female,
2. aged 18 years or older,
3. be fluent and literate in Navajo,
4. be interested and able to participate, and
5. provide written informed consent.

Exclusion Criteria:

Phase 2: History of breast cancer or mammography screening

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-03; Primary Completion 2016-07 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Acceptability of the intervention | Participants will be assesed at 3 month follow-up
  Participants will be asked if they found the intervention to be helpful or not and if they would recommend it to other women

SECONDARY OUTCOMES:
Changes in Cancer Literacy Measure | participants will be assessed at baseline and at 3 month follow-up
  Participants will be asked about breast cancer screening knowledge and attitudes including cultural barriers to screening
completion of mammography screening | participants will be assessed from the time of enrollment to 3 month follow-up
  Based on program records we will determine if participants completed mammography screening or not

CONTACTS AND LOCATIONS:
Overall Officials: Christi A Patte, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Dine College, Shiprock, New Mexico, United States